CLINICAL TRIAL: NCT03009682
Title: Phase II, Single-arm Study of Olaparib Monotherapy in Relapsed Small Cell Lung Cancer Patients With HR Pathway Gene Mutations Not Limited to BRCA 1/2 Mutations, ATM Deficiency or MRE11A Mutations(SUKSES-B)
Brief Title: Olaparib Monotherapy in Relapsed Small Cell Lung Cancer Patients With HR Pathway Gene Mutations Not Limited to BRCA 1/2 Mutations, ATM Deficiency or MRE11A Mutations
Acronym: SUKSES-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, professor, MD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-03-078
Record Dates: First submitted 2016-12-27; First posted 2017-01-04 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — olaparib

ARMS (1):
- Olaparib 300 mg (Other): Olaparib 300 mg BID per os every 12 hours administered daily. One cycle is consisted of 21 days
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Dosage and Schedule : Olaparib 300 mg BID per os every 12 hours administered daily. One cycle is consisted of 21 days.
  Two x 150 mg olaparib tablets should be taken at the same times each morning and evening of each day, approximately 12 hours apart with approximately 240 mL of water. The olaparib tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib can be taken with a light meal/snack.

SUMMARY:
This study is a single arm, multi-center phase II study of olaparib monotherapy in patients with relapsed small cell lung cancer (SCLC) harboring HR pathway gene mutations not limited to BRCA 1/2 mutations, ATM deficiency or MRE11A mutations as second or third line chemotherapy.

Target subject population:

Patients with small cell lung cancer that have progressed following first-line platinum-based therapy. Patients must have imaging confirmed progression on 1st line chemotherapy for SCLC treatment, which must have contained platinum-based regimen, with at least one measurable lesion per RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Small cell lung cancer that satisfies one or more of the following conditions:

1) BRCA1 or BRCA2 mutation, ATM deficiency, MRE11A mutation 2) Mutation of other HR(homologous recombination) pathway genes: BLM, NBN, RAD50, RAD52, RAD54L, RAD51, RAD51B, RAD51C, RAD51D, RECQL, RECQL4, RECQL5, RPA1, WRN etc.

3. Small cell lung cancer that has progressed during or after first-line therapy.

* The 1st line regimen must have contained platinum based regimen.
* Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
* If the patient correspond to sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), she/he should get second- line treatment.

  4. Patients (male/female) must be > 20 years of age.

  5. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  6. ECOG performance status 0-1 7. Patients must have a life expectancy ≥ 16 weeks 8. Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1 9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up. 10. At least one lesion, not previously irradiated, 11. Provision of informed consent for genetic research.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the last 2 weeks (or a longer period depending on the defined characteristics of the agents used).
4. Any previous treatment with a PARP inhibitor, including olaparib.
5. More than two prior chemotherapy regimen for the treatment of small cell lung cancer. Pazopanib maintenance or immune checkpoint inhibitor (CTLA4, PD-1 or PD-L1 monoclonal antibody) is not considered as line of treatment.
6. Patients with second primary cancer
7. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
8. Concomitant use of known CYP3A4 inhibitors such as ketokonazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir
9. Persistent toxicities (>=CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
10. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Patients with myelodysplastic syndrome/acute myeloid leukaemia
12. Patients with symptomatic uncontrolled brain metastases.
13. Major surgery within 14 days of starting study treatment or patients not being recovered from any effects of any major surgery
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
15. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
16. Breast feeding women
17. Immunocompromised patients,
18. Patients with known active hepatic disease (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
19. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
20. Patients with uncontrolled seizures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | Up to 30 months

SECONDARY OUTCOMES:
Duration of response | Up to 30 months
Disease control rate | at 12 weeks
Overall survival (OS) | Up to 30 months
Progression-free survival (PFS) | Up to 30 months
Number of participants with Adverse Events as Assessed by CTCAE v4.03 | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea